CLINICAL TRIAL: NCT00196989
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study of Oral GW677954 as a Monotherapy for 12 Weeks Duration in Patients With Type 2 Diabetes Mellitus
Brief Title: Study In People With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADG20001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Efficacy; PPARpan; Type 2 Diabetes Mellitus; Phase IIb; Safety; Pharmacokinetics; GW677954; Pharmacodynamics; Tolerability; Dose-Ranging
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pioglitazone
Drug: GW677954
  Other Names: Pioglitazone

SUMMARY:
This Phase 2 dose-ranging study will evaluate the efficacy, safety and tolerability of a range of doses of GW677954 compared with placebo over sixteen weeks of treatment in subjects with T2DM (Type 2 Diabetes Mellitus).

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Double-Dummy, Parallel-Group, Placebo-Controlled, Study To Evaluate Efficacy, Safety And Tolerability Of Oral GW677954 Capsules (2.5, 5, 10, 15 And 20 Mg Once A Day) As A Monotherapy (Diet and/or exercise treated) Or As An Add-On To Metformin For 16 Weeks Duration In Subjects With Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion criteria:

* Subjects with T2DM as defined by the criteria of the ADA and/or recognized by WHO Expert Committee on the Diagnosis and Classification of Diabetes Mellitus [American Diabetes Association, 2004], for at least 3 months preceding screening (see Section 15.3, Appendix 3:, "Diagnosis and Classification of Diabetes Mellitus").
* To be eligible for Randomization into the trial, a subject must satisfy all of the following glycemic criteria:

  * HbA1c level via central laboratory at the pre-screening visit
  * If HbA1c ≥ 8.0% but ≤ 10.0%: subject may proceed to Randomization;
  * If HbA1c ≥ 7.8% but < 8.0%, subject not eligible to proceed, but may be retested once to establish eligibility (or lack thereof). If HbA1c level ≥ 8.0% upon retest, subject is eligible to proceed; otherwise they should be withdrawn.
  * If HbA1c < 7.8%, subject not eligible to proceed (no retest allowed).
  * FPG level via central laboratory at the pre-screening visit must be < 270 mg/dL (15.0 mmol/L). FPG may be retested within a week to confirm eligibility (or lack thereof).
* Concurrent T2DM therapy:

  * Diet and/or exercise treated: Must not have taken antidiabetic medication for at least 2 months prior to the pre-screening visit, OR
  * Metformin monotherapy: Subjects entering the study on metformin must be on the same dose, formulation and regimen of metformin for at least 2 months prior to the pre-screening visit, AND
  * TZDs and insulin are excluded in the 3 months prior to the Screening visit for all subjects.
* Males and females who are 18 to 70 years of age inclusive at the time of Screening.
* If female, eligible to enter and participate in this study:

  * If of non-childbearing potential (i.e., physiologically incapable of becoming pregnant (tubal ligation), including any female who is post-menopausal [>1 year without menstrual period]); or,
  * If of child-bearing potential, has a negative pregnancy test at Screening (serum), at Randomization (urine) and:

    * Has a male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject, or
    * Uses double-barrier methods of contraception; condoms with the use of caps (with spermicide) and IUDs are acceptable, or
    * Uses hormonal contraceptives (oral, depots, patches etc) with double- barrier methods of contraception as outlined above, or
    * Abstains from sexual intercourse, or
    * Is with a same sex partner and does not participate in bisexual activities where there is any risk of pregnancy.
* Body Mass Index (BMI): ≥25 and ≤40 kg/m² and weigh at least 50 kg at Screening.
* If subject is a smoker, must be able to abstain while in clinic at each visit.
* Subject has given full written informed consent prior to any study related procedures are performed.

Exclusion criteria:

Exclusion Criteria:

* Metabolic Disease including:

  * Diagnosis of Type 1 diabetes mellitus
  * Uncorrected thyroid dysfunction. (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy for at least 1 month prior to Screening, and who have a screening thyroid stimulating hormone (TSH) within the upper limit of normal may participate).
  * Significant weight gain or loss (defined as > 5% of total body weight) within the 3 months prior to Screening.
* Previous use of insulin for treatment of hyperglycemia within 3 months of Screening.
* History of recent clinically significant cardiovascular disease including:

  * History or ECG evidence of prior myocardial infarction within 6 months prior to Screening.
  * Current unstable angina or history of unstable angina in past 6 months.
  * Coronary revascularization including percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) surgery that is either planned or occurred in the 6 months prior to Screening.
  * Clinically significant arrhythmia or valvular heart disease.
  * Congestive heart failure (CHF) with New York Heart Association (NYHA) Class II-IV symptoms (see Section 15.4, Appendix 4).
  * Blood pressure > 160/100 mmHg or resting heart rate > 100 bpm. Note: subjects using antihypertensives [e.g., beta blockers, angiotensin converting enzyme (ACE) inhibitors, angiotensin II antagonists, calcium channel blockers and diuretics] must be on stable doses during the 30 days prior to Screening and during the trial.
  * Has a QTc interval (Bazett's) > 440 msec in males and > 450 msec in females at Screening.
  * Clinically significant ECG abnormalities which, in the opinion of the Investigator, may affect the interpretation of safety data, or which otherwise, contraindicates participation in a clinical trial with a new chemical entity.
* History of chronic pancreatitis.
* Familial hypercholesterolemia.
* TGs ≥800 mg/dL (8.96 mmol/L) at Screening.
* Serum creatinine at screening > 1.4 mg/dL (124 µmol/L) for women, or > 1.5 mg/dL (133 µmol/L) for men.
* Clinically significant anemia defined by hemoglobin concentrations <12.0 g/dL or < 120.0 g/L for males and < 11.0 g/dL or < 110.0 g/L for females.
* History of significant co-morbid diseases (e.g., cholelithiasis, gastrointestinal disease, etc.) that would preclude participation in the study.
* Documented history of hepato-biliary disease including a history of, or positive laboratory results for hepatitis (hepatitis B surface antigen and/or hepatitis C antibody) at Screening, and/or clinically significant hepatic enzyme elevation including:

  •Any one of the following enzymes greater than 2.5 times the upper limit of normal (ULN) value at Screening:
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Alkaline phosphatase (ALP)
  * Total or direct bilirubin > 1.5 times the ULN at Screening, unless consistent with presumed or diagnosed Gilbert's disease.
* History of metabolic acidosis, rhabdomyolysis, myalgia, myositis or myopathy after taking statins or fibrates.
* Any subject who has withdrawn therapy due to AEs after taking a PPARγ or a PPARα/γ dual agonist, either marketed (e.g., troglitazone, rosiglitazone or pioglitazone) or under current or previous clinical investigation.
* Signs or symptoms of myositis at Screening (or upon 1 repeat test), and/or creatinine phosphokinase (CPK)≥3.0 times ULN
* Is currently taking or has taken any of the following medications in the 3 months prior to the pre-screening visit:

  * Anti-obesity agents (including fat absorption blocking agents)
  * St. John's Wort
  * Warfarin and other oral anticoagulants (excluding aspirin and non-steroidal anti-inflammatory drugs)
  * Digoxin
  * Oral or injectable corticosteroids (inhaled and intranasal steroids are acceptable)
  * Use of antidiabetic agents (other than metformin) in the 2 months prior to the pre-screening visit.
  * Use of TZDs in the 3 months prior to the pre-screening visit.
  * Methotrexate, cyclosporine or monoclonal antibodies (e.g., alemtuzumab, gemtuzumab ozogamicin, rituximab, trastuzumab, ibritumomab, tiuxetan) for rheumatoid arthritis or psoriasis.
  * Atypical antipsychotic medications [e.g., aripiprazole (Abilify), risperidone (Risperdal), clozapine (Clozaril), olanzapine (Zyprexa), quetiapine (Seroquel), and ziprasidone (Geodon)].
  * Antiretroviral drugs
  * Use of lipid lowering agents within 3 months prior to the pre-screening visit. This includes statins, fibrates, ezetimibe (Zetia), niacin and bile acid sequestrants.
  * Monoamine oxidase inhibitors
* History of cancer except for the following:

  * Basal cell carcinoma or superficial squamous cell carcinoma treated by local excision.
  * Cervical cancer in situ treated definitively more than 6 months prior to screening.
* Women who are lactating, pregnant, or planning to become pregnant.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to any drug chemically related to the study drug.
* Known allergy to any of the capsule excipients, or history of drug or other allergy, which, in the opinion of the responsible study physician, contradicts participation. Hypersensitivity to metformin or any of its components (for subjects entering on metformin).
* Has a history of substance and/or alcohol abuse within the past year as determined by the Investigator at screening or during treatment:

  * Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
  * History of alcohol abuse defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.
* Received treatment with a new molecular entity (investigational drug) during the previous 4 months or participated in any other trial during the previous 3 months, or has participated in a previous study with GW677954. A new molecular entity is defined as any compound not in Phase 3. (The washout is from last dose of investigational product in the previous study until the first dose of investigational product.)
* Likely to be non-compliant, in the investigator's opinion, with respect to the protocol and related scheduled visits.
* Subject has any concomitant medical condition which in the opinion of the investigator makes them unsuitable to participate in the study.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Percentage change from Baseline (Day 1) in glycated hemoglobin (HbA1c) levels at Week 16 as a measure of improvement in glucose control | Week (W) 16
  Improvement in glucose control was measured by means of reduction in glycated hemoglobin (Hb) levels in blood.

SECONDARY OUTCOMES:
Percentage change from Baseline (Day 1) in fasting HbA1c levels at Weeks 4, 8 and 12 | Weeks 4, 8, and 12
  Improvement in glucose control was measured by means of reduction in glycated hemoglobin (HbA1c) levels in blood. Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in fasting plasma glucose (FPG) at Weeks 1, 2, 4, 6, 8, 12 and 16 | W1, W2, W4, W6, W8, W12, and W16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in fasting fructosamine at Weeks 2 and 4 | Baseline (Day 1), W2, W4
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Percentage of participants achieving target HbA1c levels at Weeks 4, 8, 12, and 16 | Weeks 4, 8, 12, and 16
  Improvement in glucose control was measured by means of reduction in glycated hemoglobin (HbA1c) levels in blood. The ideal concentration of HbA1c was desired to be less than or equal to 7%.
Percentage of participants achieving a decrease in HbA1c of >= 0.7% from Baseline (Day 1) at Weeks 4, 8, 12 and 16 | Baseline (Day 1), Weeks 4, 8, 12, and 16
  Improvement in glucose control was measured by means of reduction in glycated hemoglobin (HbA1c) levels in blood.
Percentage of participants achieving target range of FPG at Weeks 1, 2, 4, 6, 8, 12 and 16 | Weeks 1,2, 4, 6, 8, 12, and 16
  The target range for FPG was <=126 milligrams per deciliter (mg/dL) or 7.0 millimoles per liter (mmol/L) to <=140 mg/dL or 7.8 mmol/L
Percentage of participants achieving a decrease from Baseline (Day 1) of >=30 mg/dL [1.66 mmol/L] in FPG at Weeks 1, 2, 4, 6, 8, 12 and 16 | Weeks 1, 2, 4, 6, 8, 12, and 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Ratio to the Baseline (percentage change) of total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), triglycerides (TG), and free fatty acids (FFA) at Weeks 2, 4, 8, 12, and 16 | Baseline (Day 1), Weeks 2, 4, 8, 12, and 16
  This data analysis was based on log-transformed data.
Percentage change from Baseline (Day 1) in non-HDL-C based on log-transformed data at Week 16 | At Week 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Percentage change from Baseline (Day 1) in very low density lipoprotein-cholesterol (VLDL-C), apolipoprotein AI (Apo AI), AII, and B at Week 16. | At Week 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in Apo B/TC, TC/HDL-C, and LDL-C/Apo B ratio at Week 16 | At Week 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in hemoglobin at Week 16 | At Week 16
  This analysis was performed in sitting position. Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in hematocrit at Week 16 | Wekk 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in systolic and diastolic blood pressure (SBP and DBP) at Week 16 | At Week 16
  Systolic blood pressure )SBP) and diastolic blood pressure (DBP) were measured in sitting position. Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in heart rate at Week 16 | Week 16
  Heart rate was measured in sitting position. Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in body weight at Week 16 | Week 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in 12 lead electrocardiogram (ECG) measures including PR interval, QT interval, QTc interval and QRS duration at Week 16 | Week 16
  QT(c) interval calculations were done by Bazett's method (QTc[B]) as well as by Fridericia's correction (QTc[F]). Change from Baseline is the value at indicated time point minus the Baseline value.
Number of participants with clinical hematology, chemistry, urinalysis, exploratory cardiac parameters of potential clinical concern (PCC) along with serum pregnancy test over period | Upto 16 weeks
  Participants were analyzed for any abnormality for laboratory parameters either higher or lower than the potential clinical concern range.
Number of participants with hypoglycemic events as a measure of ophthalmic assessment | Up to 16 weeks
  Participants received a glucose log for reading for routine recording of glucometer readings. Glucose values were recorded on timely basis.
Number of participants with intensity of hypoglycemic events as a measure of ophthalmic assessment | Up to 16 weeks
  Participants received a glucose log for reading for routine recording of glucometer readings. Glucose values were recorded on timely basis.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) over period | Up to 16 weeks
  Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Change from Baseline (Day 1) in phosphocreatine kinase (Creatine kinase-MB) over period | Up to 16 weeks
  CK-MB is a cardiac biomarker.
Number of participants with absolute Troponin-I (cTnI) levels over period | Up to 16 weeks
  Troponin-I (cTnI) is a cardiac biomarker.
Change from Baseline (Day 1) in fasting insulin at Week 8 and 16 | Week 8 and 16
  Change from Baseline is the value at indicated time point minus the value at Baseline.
Change from Baseline (Day 1) in C-peptide at Week 8 and 16 | Week 8 and 16
Change from Baseline (Day 1) in HOMA-S at Week 16 | Week 16
Change from Baseline (Day 1) in QUICKI at Week 16 | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (124):
- United States (60):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Alhambra, California
  - GSK Investigational Site, Artesia, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Inglewood, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Norwalk, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Pahrump, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Franklin, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Cite, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Monroe, Washington
  - GSK Investigational Site, Wauwatosa, Wisconsin
- Argentina (4):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, San Juan
- Australia (8):
  - GSK Investigational Site, Miranda, New South Wales
  - GSK Investigational Site, Carina Heights, Queensland
  - GSK Investigational Site, Spring Hill, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Keswick, South Australia
  - GSK Investigational Site, Port Lincoln, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
- Canada (22):
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Smiths Falls, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Granby, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Longueuil, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Bogotá, Colombia
- GSK Investigational Site, San José, Provincia de San José, Costa Rica
- Czechia (4):
  - GSK Investigational Site, Cheb
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- GSK Investigational Site, Quito, Ecuador
- Latvia (4):
  - GSK Investigational Site, Cēsis
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Tukums
- Mexico (6):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mexico City
- New Zealand (4):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Rotorua
  - GSK Investigational Site, Tauranga
- Peru (3):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Isidro, Lima region
  - GSK Investigational Site, Lima
- Russia (6):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ADG20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register